CLINICAL TRIAL: NCT03683225
Title: A Phase 2 Study to Evaluate the Safety, Tolerability and Initial Efficacy of Pramipexole ER, Given With Aprepitant in Patients With Idiopathic Parkinson's Disease
Brief Title: A Study to Evaluate in Patients With Parkinsonian Type Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chase Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTC-002
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Pramipexole ER tablets will be administered with or without aprepitant, orally once daily in the morning.
  During Part 1 and Part 2, pramipexole ER dosage will be adjusted in twice-weekly increments of 0.75 mg/day as guided by efficacy and tolerability (see table above).
  Aprepitant:
  From study Part 2 onwards, participants will also receive one 80 mg capsule of aprepitant co-administered once daily with pramipexole ER.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTC-413 (Experimental): Pramipexole with/with out aprepitant orally once daily
  Interventions: Combination Product: CTC-413

INTERVENTIONS:
Combination Product: CTC-413 — pramipexole ER, given with aprepitant

SUMMARY:
A Phase 2 study to evaluate the safety, tolerability and initial efficacy of pramipexole ER, given with aprepitant in patients with parkinsonian type disorders

DETAILED DESCRIPTION:
Methodology:

This is an initial Phase 2, rising-dose, single-blind, out-patient, sequential-treatment study in up to 24 patients with idiopathic Parkinson's disease of about 5 months duration. All participants will have idiopathic Parkinson's disease (PD).

Subjects will sign a consent form prior to any study related procedure and will complete baseline screening assessments.

The study will be conducted in three parts:

Part 1: All eligible patients switch from their dopaminergic treatment to the equivalent dose of pramipexole ER in the judgement of the investigator. Then, pramipexole ER is titrated alone up to the patients' optimal dose or to the protocol maximum allowed dose for Part 1 of 4.5 mg/day.

Part 2: Add-on aprepitant and continue the titration of pramipexole ER from the optimal dose (or 4.5 mg/day) determined in Part 1 to the optimal dose not to exceed the protocol limit of 9.0mg/day, given in combination with aprepitant.

Part 3: Maintain the dose of pramipexole ER found in Part 2 given in combination with aprepitant for 3 months with periodic safety and efficacy checks.

During Parts 1 and 2, subjects will be evaluated at in-clinic visits for safety and tolerability at intervals not to exceed once weekly ± 2 days and additionally by telephone or in-clinic visits, as considered clinically appropriate, at each dose change.

During Part 3, this optimal pramipexole ER/aprepitant regimen will be stably maintained for 3 months in association with monthly in-clinic laboratory and clinical evaluations. Safety and tolerability will continue to be evaluated by telephone or in-clinic visits, as deemed clinically appropriate.

Pramipexole ER tablets will be administered with or without aprepitant, orally once daily in the morning. Subjects will take 1-3 pramipexole ER tablets daily.

Aprepitant will be administered orally in a fixed daily dose by means of a single capsule containing 80 mg.

At study completion (or at other times in accordance with Stopping Rules given below), study medications will be discontinued, and participants will be returned to their pre-admission therapeutic regimen as considered medically appropriate. Investigators will always have the option of making necessary and appropriate changes to protocol dose optimization schedules in consultation with the Sponsor.

An independent DSMB will be appointed to have responsibility for safeguarding the interests of the trial subjects and assessing the safety and tolerability of the study treatments during the trial. The DSMB will meet when 10 patients complete the study and when all patients complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed an Institutional Review Board (IRB) approved informed consent document indicating that they understand the purpose of and procedures required by the study and are willing to participate in the study and comply with all study procedures and restrictions. Informed consent must be obtained from the patient and/or a designated representative prior to initiating screening procedures to evaluate eligibility of the study.
2. Males and females aged 40 - 80 years inclusive.
3. Meet criteria for the diagnosis of possible/ probable idiopathic Parkinson's disease (PD; Postuma RB, et al. 2015)
4. Have not previously been treated with CD/LD.
5. PD severity in the Hoehn & Yahr 2 to 3 range.

Exclusion Criteria:

1. Women who are pregnant or may become pregnant.
2. Nursing mothers.
3. Individuals who have taken a study medication (pramipexole and/or aprepitant) within 3 months of study admission.
4. Moderate and severe renal impairment (Creatinine Clearance: < 60 mL/min calculated by Cockcroft and Gault equation)
5. Severe hepatic impairment (Child-Pugh C)
6. Hypersensitivity to any component of either study medication
7. Being treated with the following medications:

   * Pramipexole
   * Centrally acting dopamine antagonists during preceding month
   * Pimozide
   * Strong CYP3A4 inducer or inhibitor
   * Warfarin (a CYP2C9 substrate)
   * Hormonal contraceptives
8. Patients considered unlikely to co-operate in the study, and/or poor compliance anticipated by the investigator.
9. Patients who have any clinically significant hypotension or ECG abnormality.
10. Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives.
11. Patients who have participated in another clinical trial with an investigational drug within previous 30 days.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events -Safety by Incidence of Treatment-Emergent Adverse Events | multiple times for the duration of the study (baseline through Month 3)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" . Incidence and nature of adverse events; vital signs;
Number of participants with change in weight | mulitple times from baseline through Month 3
  Number of participants with a change in weight (either by pounds or kilograms) from baseline
Number of participants with change in in physical examine | multiple times for the duration of the study (baseline through Month 3)
  physical examination changes General appearance,Head, eyes, ears, nose, and throat, Respiratory, Cardiovascular, Musculoskeletal, Abdomen, Neurologic, Extremities, Dermatologic, Lymphatic)
Number of participants with change in in clinical laboratory evaluations | multiple times for the duration of the study (baseline through Month 3)
  changes in clinical laboratory evaluations (Creatinine, Potassium(K+),Sodium (Na+) , Chloride (Cl-), Magnesium (Mg++), Calcium, Inorganic phosphate, Glucose, Urea,Bilirubin (Total) ,Bilirubin (direct), AST, ALT, GGT, Alkaline phosphatase, Total Protein Albumin,
Number of participants with change in Electrocardiography (ECG) | multiple times for the duration of the study (baseline through Month 3)
  ECG (standard digital 12-lead in singlicate).

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | multiple times from baseline through Month 3
  Change from baseline in the MDS-UPDRS Part 4 for motor fluctuations and dyskinesia severity will be assessed hourly x3 on assessment days.motor complications (six items). Subscale has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Total score 0-24.
modified Columbia-Suicide Severity Rating Scale | multiple times from baseline through Month 3
  3 question scale to to gage is the subject is having suicidal tendencies. If the response is "YES" to Question 1 or 2, or if the response to Question 3 reveals a concern about a significant level of suicidality, the subject would undergo a more detailed assessment by a qualified clinician who has experience in the evaluation of suicidal ideation and behavior, either at the site or by referral to an outside clinician. In either case, appropriate documentation of the clinical issues and management plan will be required in a narrative that would be placed in the subject's study record. Questions are 'yes' or 'no'
Pharmacokinetics of pramipexole and aprepitant | multiple times from baseline through Month 3
  Plasma concentrations of pramipexole and aprepitant will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Kitty Clarence-Smith, md, Study Director — KM Pharmaceutical Consulting
Locations (1):
- Quest Research, Farmington Hills, Michigan, United States